CLINICAL TRIAL: NCT06094049
Title: Evaluation of Acceptability of Folic Acid and Vitamin B12 Fortified Meals by Rural Communities of Ethiopia
Brief Title: Acceptability of Folic Acid and Vitamin B12 Fortified Meals
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Arba Minch University (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Addis Ababa University (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0137-B
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Dietary Habits
Keywords: Folic acid fortified meal; Vitamin B12 fortified meal; Preference test; Triangle test
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preference test: A preference test using a 5-unit hedonic scale will be conducted to assess the women liking of the meal prepared with fortified flour only.
  Interventions: Other: Preference test group
- Triangle test: A triangle tests will be carried out to detect any difference between the food prepared with fortified and unfortified flour.
  Interventions: Other: Triangle test group

INTERVENTIONS:
Other: Preference test group — Standard meals will be prepared including the commonly consumed porridge and/or bread using flour fortified with folic acid and vitamin B12. The meals will be prepared in the same way, by a local person who is familiar with the selected food.
  Groups: Preference test
Other: Triangle test group — Standard meals will be prepared including the commonly consumed porridge and/or bread using unfortified flour and fortified-flour with folic acid and vitamin B12. The meals will be prepared in the same way, by a local person who is familiar with the selected food and who will be blinded to the flour type.
  Groups: Triangle test

SUMMARY:
Evaluation of sensory acceptability of fortified products prior to distribution is essential. We aim to evaluate whether fortification affects sensory qualities and whether these are acceptable to rural communities. Standard meals will be prepared using unfortified and fortified-flour with folic acid and vitamin B12. Preference and triangle tests will be conducted among women residing in rural areas of Ethiopia.

DETAILED DESCRIPTION:
In Ethiopia, micronutrient deficiencies and associated morbidities remain a major public health problem that jeopardizes the development efforts of the country. Ethiopia faces a particularly high level of folate deficiency especially critical in women of reproductive age group (WRAG) (Haidar, J., 2010), which contributes to high rates of anaemia and can significantly increase the risk of Neural Tube Defects (NTDs), and neonatal and child mortality (Oumer, M., 2020; Wald, N.J., 2022). The government of Ethiopia recognizes the importance of a healthy population and thus has endorsed and implemented a number of nutrition specific and nutrition-sensitive interventions to improve the nutritional status and health of the population. Ethiopia has endorsed national multi-sectoral food and nutrition policy on November 23, 2018 to address the multifaceted nutritional problems. Ethiopia successfully implemented mandatory fortification programs for iodine, salt fortification with Iodine. More efforts and capacities are required to address similarly important and deep-rooted micronutrient deficiencies such as those of folic acid and vitamin B12. The Ministry of Health and all the health and nutrition stakeholders in Ethiopia recognize the vital importance of a preventive intervention that can reverse the current alarming rates of NTDs. Very recently, the fortification of edible oil and wheat flour with folic acid and other essential micronutrients was made mandatory in Ethiopia. However, they also are aware of the technical constraints in Ethiopia for the adoption of fortification of staple foods that are inherent in the diversity of staple foods and the scattered pattern of small mills. A large segment of vulnerable populations in Ethiopia resides in rural settings and has limited access to fortified foods in the market. Although consuming fortifiable wheat resulted in substantial decreases in the prevalence of micronutrient deficiencies in urban settings, large-scale fortified food is not a suitable approach to reaching the rural population, that depends on small scale mills for processing staple cereals such as maize, sorghum, and barley. Prior to testing the effectiveness of such intervention in improving the population health and nutrition outcomes, evaluation of the extent of sensory acceptability of the fortified products by the local community is important (Lawless et.al., 2010).

The study aims to evaluate the sensory acceptability of folic acid and vitamin B12 fortified cereal-based meals by the local communities. The evidence obtained from this trial will first provide us with a baseline understanding of potential adherence to the food made from the fortified flour, to carry on the effectiveness trial.

This study will be conducted in Arba Minch Health and Demographic Surveillance Sites (AM-HDSS) villages, Arba Minch Zuria District (AZD) and Gacho Baba District (GBD), Gamo Zone, Southern Ethiopia. The two districts have a total of 31 kebeles (the smallest administrative units in Ethiopia) with three different climatic zones, highland, midland, and lowland, among which 9 kebeles are targets of AM-HDSS, which is run by Arba Minch University. One kebele from highland and one from lowland will be selected to address the variability in food preparations techniques among kebeles of different climatic zones. To conduct the sensory acceptability test, standard meals will be prepared including the commonly consumed porridge and/or bread using unfortified flour and fortified-flour with folic acid and vitamin B12. Fortified and unfortified flour will be produced in a local meal contracted for the purpose of our project.

A preference test will be conducted among 36 WRAG using a 5-unit hedonic scale (color, test, flavor, texture/mouth feel, overall liking) with a consideration of meals prepared with fortified flour only. A triangle tests will be carried out to detect any difference between the food prepared with fortified and unfortified flour. In this test, 36 WRAG (different from the first group) will be served three bowels of the meal (one prepared from the fortified flour while the other two from non-fortified flour and vice versa) and will be asked to specify which one differs from the other two. Then if the difference is identified, the participant will be asked again to indicate whether the difference is large, medium or uncertain.

The data collection will be conducted through the combination of observation, self-administered questionnaires and interview techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (WRAG) between the ages of 15-49 years who live in households at AM-HDSS and who are:
* One or both of their parents signed an informed consent form and the girl's agreed if the participant is a teenage. A signed consent from women >19 years of age.
* Commonly participating in the food preparation
* With general good health
* Literate (able to read and write)

Exclusion Criteria:

* WRAG who are pregnant and/or are lactating
* WRAG with diagnosed/reported food allergies and food intolerances toward the prepared food

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sensory assessors (the panelists) will be WRAG, 15-49 years of age. This population group is mainly selected for this trial because: 1) the purpose of acceptability trail in this study is to test how the product will be liked by the local community, but not meant for the commercial use; 2) women's in Ethiopia are highly involved in food preparation and known to have a better understanding of meals characteristics; 2) the major target of intervention for the fortified product will be women.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women liking of the meal prepared with fortified flour only | 1 month
  In the preference test, the degree of liking of the fortified meal will be graded based on the 5 unit hedonic scale (1= dislike very much, 2=dislike slightly 3=neither like nor dislike 4=like slightly and 5=like very much).
The extent of perceived difference between fortified and unfortified flour by the women | 1 month
  Women will be served three bowels of the meal (one prepared from the fortified flour while the other two from non-fortified flour and vice versa) and will be asked to specify which one differs from the other two. Then if the difference is identified, the participant will be asked again to indicate whether the difference is large, medium or uncertain.

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, MD, PHD, Principal Investigator — University Ghent
Locations (2):
- Ethiopia (2):
  - Arba Minch Health and Demographic Surveillance System sites, Arba Minch
  - Arba Minch University, Arba Minch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haidar, J., Melaku, U. and Pobocik, R.S., 2010. Folate deficiency in women of reproductive age in nine administrative regions of Ethiopia: an emerging public health problem. South African Journal of Clinical Nutrition, 23(3), pp.132-137.
- [Background] Oumer M, Taye M, Aragie H, Tazebew A. Prevalence of Spina Bifida among Newborns in Africa: A Systematic Review and Meta-Analysis. Scientifica (Cairo). 2020 Oct 6;2020:4273510. doi: 10.1155/2020/4273510. eCollection 2020. PMID 33083093
- [Background] Wald NJ. Folic acid and neural tube defects: Discovery, debate and the need for policy change. J Med Screen. 2022 Sep;29(3):138-146. doi: 10.1177/09691413221102321. Epub 2022 Jun 23. PMID 35735352
- [Background] Lawless, Harry T., and Hildegarde Heymann. Sensory evaluation of food: principles and practices. Vol. 2. New York: Springer, 2010.
- See also: Mandatory fortification regulation endorsed by Ethiopia — https://www.thereporterethiopia.com/25738/